CLINICAL TRIAL: NCT03151018
Title: Harmonizing Optimal Strategy for Treatment of Coronary Atherosclerotic Lesions - Registry-based Study on the Effect and Safety of Onyx™, Zotarolimus-eluting Stent for Coronary Atherosclerotic Lesions: HOST-Onyx Registry
Brief Title: Effect and Efficacy of Onyx™, Zotarolimus-eluting Stent for Coronary Atherosclerosis
Acronym: HOST-ONYX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Hyo-Soo Kim, Professor, Seoul National University Hospital
Other Study IDs: HOST-ONYX
Record Dates: First submitted 2016-07-21; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome; Myocardial Infarction; Angina Pectoris
Keywords: coronary artery disease; percutaneous coronary intervention; zotarolimus-eluting stents
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Myocardial Infarction; Angina Pectoris

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Onyx: The patients who received PCI with Resolute Onyx stent(s)
  Interventions: Device: Resolute Onyx

INTERVENTIONS:
Device: Resolute Onyx
  Other Names: Zotarolimus-eluting stent

SUMMARY:
The objectives of this study are

1. To establish a prospective registry of the whole patients who received percutaneous coronary intervention with Resolute Onyx™ stent.
2. To evaluate the long-term efficacy and safety of coronary stenting with the Resolute Onyx™ stent.
3. To compare the long-term efficacy and safety of coronary stenting between the Resolute Onyx™ stent and other contemporary drug-eluting stents which had established their own registry.

DETAILED DESCRIPTION:
Secondary endpoints are

1. Stent thrombosis-24 hours(acute), 30 days(subacute), 1 year(late), every 1 year till 3 years(very-late) after index PCI (percutaneous coronary intervention),
2. Target vessel failure
3. Composite rate of cardiac death and any MI, 3 years
4. Composite rate of all death and any MI
5. Composite rate of all death, any MI, and any repeat revascularization
6. Compliance and therapy interruptions with prescribed adjunctive antiplatelet therapy
7. Clinical device and procedural success

ELIGIBILITY:
Inclusion Criteria:

* Age above 19
* Patients who received PCI with Resolute Onyx™ stent(s)

Exclusion Criteria:

* None

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All coronary arterial disease patients who received percutaneous coronary intervention with Resolute Onyx™ stent(s)
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure | 12 months
  Composite of cardiac death, non-fatal target vessel-related myocardial infarction (MI), and ischemia-driven target lesion revascularization (TLR)

SECONDARY OUTCOMES:
Stent thrombosis, acute | within 24 hours after index PCI
  according to Academic Research Consortium (ARC) definition
Stent thrombosis, subacute | from 24 hours to 30 days after index PCI
  according to ARC definition
Stent thrombosis, late | from 30 days to 1 year after index PCI
  according to ARC definition
Stent thrombosis, very-late | 1 year ~ up to 3 years
  according to ARC definition
Target vessel failure | 12 months
  Composite of cardiac death, non-fatal target vessel related myocardial infarction, and ischemia-driven target vessel revascularization (TVR)
Composite rate of cardiac death and myocardial infarction | 12 months, 3 years
  as title
Composite rate of all-cause death and any myocardial infarction | 12 months, 3 years
  as title
Composite rate of all-cause death and any myocardial infarction, and any repeat revascularization | 12 months, 3 years
  as title
Rate of compliance and interruptions with prescribed adjunctive antiplatelet therapy | 12 months, 3 years
  we will estimate this outcome with relevant questionnaire
Clinical device and procedural success rate | intraoperative ( index PCI)
  device success : residual stenosis <30%, final thrombolysis in myocardial infarction (TIMI) flow grade III procedural success : device success + no adverse events immediate after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-soo Kim, MD, PhD, Study Chair — Seoul National University Hospital
Locations (16):
- South Korea (16):
  - Kosin University Gospel Hospital, Busan
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Myongji Hospital, Goyang
  - Gwangju Christian Hospital, Gwangju
  - Kwangju Veterans Hospital, Gwangju
  - Chungbuk National University Hospital, Jeonju
  - Presbyterian Medical Center, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Pusan National University Hospital, Pusan
  - Seoul National University Bundang Hospital, Seongnam
  - Gangbuk Samsung Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Soonchunhyang University Hospital, Seoul
  - St. Vincent's Hospital, Suwon